CLINICAL TRIAL: NCT06621160
Title: Investigation of Spinal Posture and Anthropometric Characteristics of Women with Chronic Constipation
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Deniz Çakır, Principal Investigator, Ondokuz Mayıs University
Other Study IDs: 16/2022
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Chronic Constipation
Keywords: Chronic Constipation; Posture; Anthropometric Measurement; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: The control group consists of healthy women.
  Interventions: Other: Observation
- CC Group: The CC group consists of women with chronic constipation.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — After the participants' physical and sociodemographic characteristics were recorded, they were asked to fill out the Constipation Severity Scale and 7- Day Stool Diary to determine their constipation levels. The individuals' anthropometric characteristics were assessed with triceps, subscapula, suprailiac and calf skinfold thickness, humerus and femur epicondyle diameter, biceps and calf circumference measurements, spinal postures were assessed with the Spinal Mouse, and physical activity levels were assessed with the International Physical Activity Questionnaire-Short Form UFAA-KF and pedometer.

SUMMARY:
The aim of this study was to compare the spinal posture and anthropometric characteristics of women with Chronic Constipation (CC) and healthy women.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for women with chronic constipation:

  * Constipation according to Rome IV criteria between the ages of 18-65
  * Volunteer
  * Literacy
* Inclusion criteria for healthy women:

  * No constipation according to Rome IV criteria between the ages of 18-65
  * Volunteer
  * Literacy

Exclusion Criteria:

* Cancer, neurological disease, serious or uncontrolled systemic or metabolic disease

  * Being pregnant
  * Having a mental problem that will prevent cooperation
  * Having alarm symptoms over the age of 50
  * Having a diagnosis of secondary constipation
  * Being BMI>35
  * Having megacolon/megarectum and inactive (lazy) bowel syndrome
  * Having had colostomy surgery
  * Having a history of recent abdominal surgery
  * Having an open wound or local tumor in the abdominal region
  * Having an abdominal hernia

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: women with and without chronic constipation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Anthropometric Characteristics | 1 year
  The individuals anthropometric characteristics were assessed with triceps, subscapula, suprailiac and calf skinfold thickness, humerus and femur epicondyle diameter, biceps and calf circumference measurements.
  Triceps skinfold thickness, subscapula skinfold thickness, suprailiac skinfold thickness, calf skinfold thickness were measured with skinfold caliper; humeral epicondyle diameter, femoral epicondyle diameter were measured with mechanical caliper, biceps circumference, calf circumference were measured with tape measure. Skinfold thickness measurements were performed by the same person. The measurements were taken from the dominant side of the individuals. The measurements were performed on healthy skin and the areas to be measured were marked with a marker. The individuals were asked to relax their muscles while the measurement was performed. The skin in the marked areas was pulled up by pinching between the index finger and thumb, and the skinfold caliper was placed 1 cm below t
Spinal Posture | 1 year
  The individuals spinal postures were assessed with the Spinal Mouse. Individuals were informed about the device used and the duration of the assessment. Before the measurement, the positions in which the assessment would be made and how to do these positions were explained to the individuals. Then, a trial measurement was made once. The individuals' demographic information was entered into the computer software. Individuals were asked to stand symmetrically with their vertebral columns exposed, to take off their shoes and step onto the mat, and to distribute their weight equally on both feet on a flat surface. Spinal processes starting from C7 to S3 were determined by the physiotherapist and marked with a felt-tip pen. For measurements, the Spinal Mouse device was moved from C7 to the S3 spinous process.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant İzzet Baysal University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No